CLINICAL TRIAL: NCT06839092
Title: Prophylactic PIPAC for Reducing the Risk of Peritoneal Carcinomatosis in Patients With Colorectal Cancer: the PROPAC Randomized Clinical Trial
Brief Title: Prophylactic PIPAC in Patients With High-risk Colorectal Cancer
Acronym: PROPAC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jeremy Meyer (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Jeremy Meyer, Dr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROPAC
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer Control and Prevention; Colorectal Cancer; Colorectal Cancer Stage II; Colorectal Cancer Stage III
Keywords: Colorectal cancer; Peritoneal carcinomatosis; PIPAC; Pressurized intraperitoneal aerosol chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prophylactic PIPAC (Experimental): Standard surgery (consisting in removal of the primary cancer) followed by 6 months of adjuvant chemotherapy associated with 3 cycles of oxaliplatin-based PIPAC (4-6 weeks apart).
  Interventions: Procedure: oxaliplatin-based PIPAC
- No prophylactic PIPAC (Active Comparator): Standard surgery followed by 6 months of adjuvant systemic chemotherapy.
  Interventions: Procedure: Control (Standard treatment)

INTERVENTIONS:
Procedure: oxaliplatin-based PIPAC — Patients operated for pT4 pN0-2 cM0 pMMR colorectal cancer (of the colon, colorectal junction or high rectum) or patients operated for pT3-4 pN0-2 cM0 pMMR colorectal cancer with positive cytology or in patients with pT3-4 pN0-2 M1c pMMR colorectal cancer with limited peritoneal carcinomatosis which is limited to one abdominal quadrant and was resected during index surgery and no other distant lesion, will undergo 6 months of adjuvant systemic chemotherapy associated with 3 cycles of oxaliplatin-based PIPAC (4-6 weeks apart).
  Each PIPAC session will include exploration laparoscopy (with PCI score), peritoneal lavage for cytology and biopsies of healthy peritoneum of the four quadrants + Douglas + omentum), and oxaliplatin-based PIPAC.
  Arms: Prophylactic PIPAC
Procedure: Control (Standard treatment) — Patients operated for pT4 pN0-2 cM0 pMMR colorectal cancer (of the colon, colorectal junction or high rectum) or patients operated for pT3-4 pN0-2 cM0 pMMR colorectal cancer with positive cytology or in patients with pT3-4 pN0-2 M1c pMMR colorectal cancer with limited peritoneal carcinomatosis which is limited to one abdominal quadrant and was resected during index surgery and no other distant lesion, will undergo 6 months of adjuvant systemic chemotherapy, followed by exploration laparoscopy (including 300ml peritoneal lavage for cytology and seven punch peritoneal biopsies in the four quadrants of the abdomen, Douglas and omentum, as well as peritonectomy of 1 cm2) at 6 months after index surgery before entering a standard surveillance program.
  Arms: No prophylactic PIPAC

SUMMARY:
In a multicentric randomized controlled trial, we will compare standard surgery (consisting in removal of the primary cancer) followed by 6 months of adjuvant chemotherapy associated with 3 cycles of oxaliplatin-based PIPAC (4-6 weeks apart), to standard surgery followed by 6 months of adjuvant systemic chemotherapy (routine treatment), in patients with colorectal cancer at high risk for metachronous peritoneal carcinomatosis (pT4 pN0-2 cM0 pMMR colorectal cancer of the colon, colorectal junction or high rectum and/or with positive cytology) in terms of 1-year and 3-year peritoneal metastasis-free survival (as measured by imaging and/or surgical exploration), 1-year and 3-year disease-free survival, as well as 1-year and 3-year overall survival. In terms of outcomes measurement, patients in both groups will benefit from diagnostic laparoscopy at 6 months from the index surgery, and standard surveillance consisting in clinical examination, CEA determination and thoraco-abdominal CT at 6, 12, 24, 36, 48 and 60 months after index surgery.

ELIGIBILITY:
Inclusion criteria:

* Patients operated (in emergency or elective settings) for colorectal cancer (of the colon, colorectal junction or high rectum).
* Definitive pathological stage pT4 pN0-2 cM0 pMMR and/or pT3-4 pN0-2 cM0 pMMR with positive cytology and/or pT3-4 pN0-2 M1c pMMR with limited peritoneal carcinomatosis which is limited to one abdominal quadrant and was resected during index surgery and no other distant lesion (small indeterminate pulmonary nodules to be followed are accepted)
* Performance status 0-1.
* Age > 18 years.
* Written informed consent.

Exclusion criteria:

* Infraperitoneal rectal cancer (middle or low rectum).
* Age <18 year old.
* Age > 80 year old.
* Hereditary colorectal cancer.
* dMMR/MSI colorectal cancer.
* Inflammatory bowel disease.
* Distant metastasis (outside limited peritoneal carcinomatosis which is limited to one abdominal quadrant and was resected during index surgery and no other distant lesion; small indeterminate pulmonary nodules to be followed are accepted)
* Neo-adjuvant treatment.
* Pregnancy or lactation.
* Immunosuppression.
* Unable to provide informed consent.
* Previous cytoreductive surgery (CRS) (outside limited resection of peritoneal carcinomatosis during index surgery).
* Contraindication to laparoscopy (e.g. severe adhesions, peritonitis).
* Contraindication to and/or no adjuvant chemotherapy.
* History of allergic reaction to oxaliplatin or other platinum-containing compounds.
* Renal impairment, defined as GFR < 50 ml/min, (Cockcroft-Gault equation).
* Myocardial insufficiency, defined as NYHA class > 2.
* Impaired liver function defined as bilirubin ≥ 1.5 x UNL (upper normal limit).
* Inadequate hematological function defined as ANC ≤ 1.5 x 109/l and platelets ≤ 100 x 109/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
1-year peritoneal metastasis-free survival, | 1-year
  The primary endpoint will be the 1-year peritoneal metastasis-free survival, defined as the absence of peritoneal carcinomatosis at 1 year after index surgery, as determined during surveillance. Peritoneal carcinomatosis can diagnosed by any existing modality (as part of a pragmatic approach), including imaging (practiced during surveillance and/or in emergency for ex. for bowel occlusion), surgical exploration (practiced during PIPAC sessions in the intervention group, but also at 6 months after index surgery in the control group, which decrease the risk potential detection bias) and/or pathology. Positive cytology during exploration laparoscopy performed during PIPAC session and/or in the control group will be considered as peritoneal metastasis and therefore as a positive primary outcome.

SECONDARY OUTCOMES:
3-year peritoneal metastasis-free survival | 3-year
Disease-free survival (DFS) | 1-year, 3-years
Overall survival (OS) | 1-year, 3-year
30-day incidence of complications | 30-day
EORTC QLQ-C30 score 29 | 1 month, 2 months, 4 months, 6 months, 12 months, 24 months and 36 months

IPD SHARING:
Plan to Share IPD: Undecided